CLINICAL TRIAL: NCT04248985
Title: Effect of Bedside Ultrasound Pre-imaging on CPR Pauses in Out of Hospital Arrest
Brief Title: Effect of Pre-imaging on Cardiopulmonary Resuscitation (CPR) Pause
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Romolo Gaspari, Principal Investigator, University of Massachusetts, Worcester
Other Study IDs: UMASS-CPR2019
Record Dates: First submitted 2020-01-24; First posted 2020-01-30 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2020-07

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Intervention: Baseline measurement of timing and behavior in OOH cardiac arrest patients presenting with ongoing CPR.
  Interventions: Other: Pre-Imaging - an ultrasound technique of acquiring images
- Post-Intervention: Timing and behavior in OOH cardiac arrest patents presenting with ongoing CPR
  Interventions: Other: Pre-Imaging - an ultrasound technique of acquiring images

INTERVENTIONS:
Other: Pre-Imaging - an ultrasound technique of acquiring images — Technique involves finding low quality images of the heart during CPR prior to pausing CPR to acquire high quality images once CPR is paused.

SUMMARY:
Patients presenting following out of hospital cardiac arrest will undergo bedside ultrasound as per the hospital clinical practice. Initial 6 months include recording of current state of practice and timing of pauses and timing of ultrasounds. The second 6 months will follow an educational intervention to teach "pre-imaging". This is the technique of imaging the heart during cardiopulmonary resuscitation (CPR) to find the heart and center it on the ultrasound screen before CPR is stopped. The goal is to decrease CPR pause times when ultrasound is performed post out of hospital (OOH) cardiac arrest.

DETAILED DESCRIPTION:
There are two educational Interventions where residents will be trained in how to improve on sonographic imaging techniques performed during resuscitation following cardiac arrest. The two techniques are 1) Sonographic Pre-Imaging and 2) Sonographic Pulse Checks.

Sonographic pre-imaging Sonographic pre-Imaging involves identification of minimal cardiac details when CPR is ongoing. It involves placing the ultrasound transducer on the epigastric region during CPR to identify the general location of the heart and to center the heart in the screen prior to the point when CPR is halted. Pre-imaging produces images of the heart that insufficient for diagnostic evaluation, but allows the clinician to be in place once CPR is halted to obtain higher quality images rapidly.

Residents will be filmed during the resuscitation using two digital video cameras mounted in the resuscitation bay in the Emergency Department. One camera will be isolated to the cardiac monitor display. The other camera will be focused on the area of the room where CPR is performed. The view of this camera will focus on the torso of the patient where CPR and ultrasound imaging occurs. The camera is located in an area of the emergency department where only the patient undergoing resuscitation will be imaged. Filming will be reviewed the following day to record timing measurements of CPR and information on cardiac rhythm during CPR. All video images will be deleted within 3 days of recording to allow for recording over the weekends. No images will be saved.

The study will have three Phases.

Phase 1 - Baseline measurements of CPR activity Residents overseeing resuscitation efforts post-cardiac arrest will be eligible for inclusion in the study when providing care for patients experiencing an out-of-hospital cardiac arrest requiring resuscitation at the University Campus Emergency Department. Education on advanced cardiac life support (ACLS) is standardized through participation in an ACLS training program. A review of ACLS protocols and additional education on the importance of limiting pauses during CPR will be provided to all residents in the residency prior to initialing the study.

Medical records and video recordings will provide information on 1) Patient demographics 2) Resuscitation Interventions 3) Ultrasound Imaging 3) Timing of CPR 4) Cardiac Rhythm. Information on the actions during pauses in CPR will be used to categorize each pause. Pulse Check Pauses are occurrences when CPR is halted to feel for the presence of any pulse. Rhythm Check Pauses are occurrences when CPR is halted to determine the underlying cardiac rhythm. Defibrillation Pauses are occurrences when CPR is halted to deliver defibrillation. Vascular Access Pauses are occurrences when CPR is halted to facility the placement of central or peripheral vascular access. Airway Pauses are occurrences when CPR is halted to facilitate placement of an airway device or check the location of an airway device. Ultrasound Pauses are occurrences when CPR is halted to facilitate ultrasound imaging of the heart. Medication Pauses occur when CPR is halted to deliver intravenous or intra-osseous medications. Rhythm Change Pauses occur when CPR is halted due to a change in rhythm that does not require CPR. Patients may have pauses that involve more than one category, or no pauses at all. Summarized in Table below

Categories of Pauses in CPR Action Occurring During Pause

1. - Pulse Check Pauses Palpation for pulse in groin or neck
2. - Rhythm Check Pauses Interpret rhythm on monitor
3. - Defibrillation Pauses Defibrillate patient
4. - Vascular Access Pauses Insert peripheral or central vascular access
5. - Airway Pauses Insert of check location of airway device
6. - Ultrasound Pauses Obtain ultrasound images of heart
7. - Medication Pauses Administer medication
8. - Rhythm Change Pauses Change in rhythm resulting in no need for CPR

   Primary outcome will be the length and number of pauses in CPR during resuscitation. Measurements will be standardized by length of resuscitation (time patient arrives in emergency department to time resuscitation efforts halted) and multivariate logistic regression will be used to control for variability between patients.

   Phase 2 - Ultrasound Education Phase - Pre-imaging Education Similar to phase one, Residents overseeing resuscitation efforts post-cardiac arrest will be eligible for inclusion in the study when providing care for patients experiencing an out-of-hospital cardiac arrest requiring resuscitation at the University Campus Emergency Department. Residents will undergo standardized training on sonographic pre-imaging prior to participation in the study. They will be instructed on how to obtain pre-images and how to record images as quickly as possible during pauses in CPR. All measurements and recordings during phase 2 will be identical to phase 1. All other methodologies will remain unchanged. Primary outcome will be the length and number of pauses in CPR during resuscitation.

   All measurements and recordings during phase 1 and 2 and all other study methodology will be identical to phases 1 and 2. All other methodologies will remain unchanged.

   b. Inclusion/Exclusion Criteria - As appropriate, explain what steps will be taken to insure that subjects meet the criteria (e.g. healthy, not pregnant, etc).

   Inclusion Residents who have consented to the study will be included during episodes when a patient presents to the Emergency Department in Cardiac Arrest receiving ACLS in the Emergency Department

   Exclusion
   * Residents who do not consent to the study
   * Residents episodes where resuscitation efforts are terminated due to end of life decisions
   * Residents episodes involving the resuscitation of a trauma patient
   * Residents episodes involving patient who are not imaged with ultrasound during the resuscitation

     c. Discuss the number of experimental and control subjects, and explain the statistical basis for the numbers.

   There is limited data on pauses during CPR in the emergency department. We assumed that pauses in CPR average 15 seconds based on clinical experience. For the purpose of a power calculation, we assumed that education on pre-imaging will decrease pauses during ultrasound imaging by 5 seconds and imaging in the groin will decrease pauses by 10 seconds. Assuming an 80% power and an alpha of 0.05 we need 79 patients in phase one and 63 patients in phase two and 16 patients in phase three. Because of clustering around individual providers we will need to enroll two times that amount be account for clustering by provider. This means we need to enroll a total of 300 patients.

   Phase 3 -

   Sonographic Pulse Checks - Exploring the use of doppler imaging of the femoral artery during and between CPR to replace palpation of the pulse.

   Similar to phases one and two, residents overseeing resuscitation efforts post-cardiac arrest will be eligible to participate in the study when providing care for patients experiencing an out-of-hospital cardiac arrest requiring resuscitation at the Emergency Department. Clinicians or research staff will perform sonographic pulse checks by imaging the femoral or cardiac artery and visualize any flow within the vessel. Sonographic pulse checks will occur either a) during CPR b) during pauses in CPR c) during transitions from CPR to pause or d) during transition from pause to CPR.

   Patient inclusion and exclusion criteria are identical to phase 1 and 2.

   Patients will undergo standard of care as per UMass practice. This includes ACLS interventions based on published ACLS protocols. During pauses in CPR clinicians perform brief echocardiography of the heart, with attention to not delaying CPR pauses. During the same pause doppler imaging of the CFV will be performed by research or clinical staff. Clips of any of the 4 time periods listed above will be digitally recorded. Simultaneous clips of the patients heart will be digitally recorded.

   Patients will be followed to survival endpoints including a) ROSC b) survival to hospital admission c) survival to hospital discharge and d) death in ED. Survival endpoints will be abstracted from the medical record.

   Digital images will be de-identified and paired by patient and pause. (Patient X, pause 1; Patient X, pause 2...). Interpretation of the brief echo will be to identify the presence or absence of cardiac activity and to identify if the cardiac activity is organized or not. In addition, the images will be reviewed to identify ventricular fibrillation. Interpretation of the CVF doppler images will be performed to identify a) VTI and maximal velocity of arterial pulses from CPR b) VTI and maximal velocities of arterial pulses secondary to cardiac activity c) Rate and regularity of CPR pulses, d) rate and regularity of cardiac activity pulses e) inherent noise level of doppler signal between pulses.

   This is a proof-of-concept, descriptive study without a specific power analysis. The goal is to describe the amount of cardiac activity as visualize during brief echo that corresponds to measurable pulse activity by doppler. The secondary goal is to determine if the presence of an "irregular pulse" during regular CPR is associated with ROSC.

ELIGIBILITY:
Inclusion Criteria:

* Atruamatic Out of hospital Cardiac Arrest

Exclusion Criteria:

* physician not credentialed in bedside ultrasound
* video images not recorded (lost data)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient presenting to the emergency department in Out of Hospital Cardiac Arrest
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Length of CPR pause | 1 year
  the time between stopping CPR and restoring CPR during resuscitation.

SECONDARY OUTCOMES:
Survival | 1 year
  survival to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Romolo Gaspari, MD, PhD, Principal Investigator — UMass Worcester
Locations (1):
- UMASS Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gaspari RJ, Lindsay R, Dowd A, Gleeson T. Femoral Arterial Doppler Use During Active Cardiopulmonary Resuscitation. Ann Emerg Med. 2023 May;81(5):523-531. doi: 10.1016/j.annemergmed.2022.12.002. Epub 2023 Feb 7. PMID 36754697